CLINICAL TRIAL: NCT03875261
Title: Effect of Cannabinoid (THC / CBD 50%) on Hyperalgesia in Patients With Deep Endometriosis
Acronym: EdomTHC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: David Garcia Cinca (Other)
Collaborators: Fundació Clínic per la Recerca Biomedica (Unknown); Dr. Christian Dursteler (Unknown)
Responsible Party: Sponsor-Investigator, David Garcia Cinca, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004378-92
Record Dates: First submitted 2019-03-06; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Participants are treated with the investigational medical product
  Interventions: Drug: Cannabinoid treatment

INTERVENTIONS:
Drug: Cannabinoid treatment — Participants are treated with cannabinoid derivates with a dose between 1 to 12 puffs, each puffs contains 2,7 mg of delta-9-tetrahidrocannabinol and 2,5 mg of cannabidiol.

SUMMARY:
This study evaluates the treatment of the symptoms of deep endometriosis with a cannabinoid derivate.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 40.
* Diagnosis of deep endometriosis after clinical suspicion and confirmation by imaging test.
* Pain with a score of 4 or more on a numerical visual scale of 11 levels (EVN 0-10) in the last 3 months (includes any type of pain associated with endometriosis: dysmenorrhea, dyspareunia, dyschezia, dysuria and / or pelvic pain).
* Women of childbearing age * should have a negative pregnancy test before inclusion in the study and should commit to using highly effective contraceptive methods (hormonal contraceptives, intrauterine device, intrauterine hormonal release systems, bilateral tubal occlusion, vasectomy the couple, barrier methods and sexual abstinence) during the entire duration of the study and up to 3 months after the end of it.
* Acceptance of participation in the study by signing the informed consent.

Exclusion Criteria:

* Patients previously submitted to open abdominal surgery.
* History of cancer.
* Suspicion or diagnosis of endocrine, cardio-vascular or systemic pathology relevant.
* Pregnancy or anticipation of pregnancy up to 3 months after the end of the study.
* Current breastfeeding.
* Use of hormonal treatment (combined oral contraception, progestin in the 3 months prior to the study, GNRH analogs in the 6 months prior to the start of the study).
* Use of other analgesics different from those allowed in the study.
* Recreational or pharmacological use of cannabinoids.
* Hypersensitivity to cannabinoids or any of the exceptions.
* Known or suspected personal history, or family history of schizophrenia or other psychotic illnesses, severe personality disorder or other major psychiatric disorders.
* Patients with liver or kidney failure, severe cardiovascular disease and a history of epilepsy or recurrent seizures.
* Patients who use concomitant potent enzyme inducers of CYP3A4, such as rifampicin, carbamazepine, phenytoin, phenobarbital, and St. John's wort.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Pressure threshold in hypogastrium that induces pain | day 30 after treatment initiation
  Pain threshold versus mechanical stimulation in hypogastrium (anterior central L2 dermatoma) measured in kPa

SECONDARY OUTCOMES:
Pressure threshold in dermatomes that induces pain | baseline, day 15, day 30 and day 45
  Umbral of pain versus mechanical stimulation in dermatomes L2 anterior, L2 posterior, and T1 of the dominant upper extremity.
Temperature threshold in dermatomes that induces pain | baseline, day 15, day 30 and day 45
  Umbral sensation versus thermal stimulus (cold heat) in anterior central L2 dermatomes, posterior central L2, and T1 of the dominant upper extremity. Measured in ºC.
Intensity of the general pain | baseline, day 15, day 30 and day 45
  Intensity of the general pain associated with endometriosis measured by a visual analogue scale (0-10)
Anxiety and depression combined scale | baseline, day 15, day 30 and day 45
  Anxiety and depression measured with the Scale of Anxiety and Hospital Depression Scale (HADS).
Quality of Life | baseline, day 15, day 30 and day 45
  Quality of Life measured through the EQ-5D-5L questionnaire.
Central sensitivity | baseline, day 15, day 30 and day 45
  Central sensitivity measured with the Central Sensitization Inventory (CSI) questionnaire.
Cognitive disorder measured by a list of words | baseline, day 15, day 30 and day 45
  Cognitive disorder measured by a list of words (immediate memory and retention) and digits (attentional capacity) of the Wechsler Memory Scale (WMS-III).
about sleep quality | baseline, day 15, day 30 and day 45
  Visual analogue scale 0-10 about sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain